CLINICAL TRIAL: NCT07239882
Title: The Effect of a Digital Board Game-Based Psychological Empowerment Program on Nurses' Psychological Empowerment Levels, Job Satisfaction, and Innovative Behaviors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, MERVE OZLU, Doctoral student, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1225794
Record Dates: First submitted 2025-07-31; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Digital Board Games; Intervention; Psychological Empowerment Program
Keywords: Nursing; Psychological Empowerment; Job Satisfaction; Digital Board Games; Innovative Behavior; intervention

STUDY DESIGN:
Intervention Model Description: "The intervention group will participate in 6 weekly sessions, each consisting of a 1-hour online educational presentation and a 1-hour online group workshop using digital board games. The program is designed to last 6 weeks, and follow-up assessments will be conducted 1 and 3 months after completion to evaluate sustainability of effects. The control group will not receive active intervention during the study but will be provided with the educational booklet at the end. Both groups will be assessed at the same time intervals."
Who Masked: Outcomes Assessor
Masking Description: "Randomization will be performed by an independent researcher. Group allocation will not be revealed to the data analyst during statistical evaluation."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Board Game-Based Psychological Empowerment Program (Experimental): Nurses in the intervention group will participate in a 2-hour online psychological empowerment program, once a week for 6 weeks. The program will consist of online educational presentations, group discussions, digital board game activities (via the Board Game Arena platform), and session evaluations conducted using the Kahoot application. The program aims to increase nurses' psychological empowerment, improve their job satisfaction, and support their innovative behaviors. Sustainability assessments will be repeated 1 month and 3 months after the intervention.
  Interventions: Behavioral: Digital Board Game-Based Psychological Empowerment Program
- Control Group - Standard Application (No Intervention): Nurses in the control group will not receive any active intervention. However, they will be provided with a booklet version of the psychological empowerment program training content after the study is completed. Pretests, posttests, and follow-up measurements (months 1 and 3) will also be administered at the same time as the intervention group.

INTERVENTIONS:
Behavioral: Digital Board Game-Based Psychological Empowerment Program — This intervention is a 6-week online program aimed at increasing nurses' psychological empowerment, job satisfaction, and innovative behavior. Each session will last 2 hours and will be conducted via Zoom. The program will consist of:
  Online educational presentations on psychological empowerment, Group discussions and experience sharing, Digital board games via the Board Game Arena (BGA) platform, Session evaluations using the Kahoot app (increasing motivation by offering small prizes to the first 3 participants).
  The intervention group will receive a pretest, posttest, and sustainability measurements (1- and 3-month follow-ups).
  Arms: Digital Board Game-Based Psychological Empowerment Program

SUMMARY:
Psychological empowerment is defined as nurses' perceptions of their professional roles as meaningful, their ability to effectively perform their duties, their level of participation in organizational decision-making processes, and their perceptions of their professional productivity. In occupational groups with high stress levels, such as nursing, psychological empowerment plays a crucial role in maintaining individual and organizational well-being. Research indicates that nurses' levels of psychological empowerment are moderate and that there is a need for enhancing interventions.

The purpose of this study is to evaluate the effects of a digital board game-based psychological empowerment program on nurses' psychological empowerment levels, job satisfaction, and innovative behaviors. The research was designed with a pretest-posttest randomized controlled experimental design. The study sample will consist of nurses working in a university hospital. Participants will be selected according to specified inclusion and exclusion criteria, and data will be collected using a Personal Information Form, the Psychological Empowerment Scale, the Job Satisfaction Scale, and the Innovative Behavior Scale. The "digital board game-based psychological empowerment program" will be structured based on Kanter and Spreitzer's empowerment theories. The Ministry of Health's 2021 "Guide to Core Competencies in Nursing," the Psychological Empowerment Scale sub-dimensions, and studies on psychological empowerment in nursing in the literature will be considered in the preparation of the training content. The final version of the program will be completed following expert opinions. The program will consist of 6-week sessions. Each session is planned as two parts: (1) online empowerment training and (2) online group workshops. The group workshops will include topic-specific question-and-answer activities, group discussions, and digital board game applications appropriate to the session theme. Re-measurements (post-tests) will be conducted in the first and third months following the intervention. The control group will not receive any active intervention and will be subjected to the same assessment at the same time intervals as the intervention group. The control group will receive a booklet containing the training content at the end of the study. The data obtained will be analyzed using an independent samples t-test. The study results indicate a significant increase in nurses' psychological empowerment levels and an improvement in their job satisfaction and innovative behaviors in the intervention group. While numerous studies on the psychological empowerment of nurses exist in the literature, structured, long-term psychological empowerment programs and intervention studies are limited. The unique aspect of this study is the development and implementation of an innovative game-based intervention program to contribute to the psychological empowerment of nurses.

DETAILED DESCRIPTION:
Benner defines power as the caring practices nurses use to empower their patients. In nursing theories, the concept of "power" is emphasized as the nurse's ability to influence patients, their families, colleagues, and their work in general. The challenges nurses face and the inadequate recognition of their sources of power lead them to feel powerless, ineffective, and undervalued . Negative outcomes such as job dissatisfaction, burnout, and poor professional performance are observed in nurses who experience a sense of powerlessness. Empowerment is defined as granting appropriate responsibilities, increased authority, and authority to employees. Empowerment is known to occur at both structural and psychological levels. Psychological empowerment is generally not dependent on managerial practices but is related to how employees perceive these practices and aims to increase an individual's motivation towards their work, foster ownership of their work, and strengthen decision-making ability. Psychological empowerment consists of four main dimensions: meaning, competence, autonomy, and impact.

* Meaning: The alignment of a job with an individual's beliefs, values, and behaviors.
* Competence: The belief that an individual can perform their job effectively.
* Autonomy: The employee's freedom and control over how their job is performed.
* Impact: The employee's sense of being able to influence strategic and organizational outcomes in the workplace.

Empowered nurses perform their professional roles more effectively and improve the quality of patient care. In occupational groups with high stress levels, such as nursing, psychological empowerment plays a crucial role in maintaining individual and organizational well-being. It is known that research on nursing empowerment focuses primarily on activities that increase structural empowerment. However, in some cases, institutional and environmental arrangements for structural empowerment are not sufficient for nurses' empowerment. In such cases, it may be more beneficial for nurses to psychologically empower themselves and their teammates. Furthermore, the fact that empowerment only works when employees feel empowered increases the importance of psychological empowerment. The literature has reported that factors such as challenging working conditions and a lack of resources, information, and support in the work environment affect psychological empowerment. Nurses' levels of psychological empowerment are also influenced by organizational structure, leadership style, communication style, participation in decision-making, and professional development opportunities. According to self-efficacy theory, an individual's belief in their own abilities and their success experiences in their professional lives are also determining factors in the development of their sense of empowerment. Studies have revealed that nurses' psychological empowerment levels are moderate and this status demonstrates significant relationships with job satisfaction, burnout, motivation, and innovative behaviors. Ensuring nurses' psychological empowerment and job satisfaction is vital for achieving better health outcomes, improving the quality of care and patient safety, reducing nurse turnover, and ensuring the sustainability of global health systems.

Empowerment not only increases nurses' commitment to their work but also reduces perceptions of burnout, increases job satisfaction and productivity, and improves the quality of healthcare. Feeling empowered is critical for nurses' adaptability to innovation, leadership skills, and successful work outcomes. However, unmeasured productivity, negative attitudes, and inadequate administrative support lead to a sense of powerlessness among nurses. Therefore, initiatives aimed at increasing their levels of psychological empowerment are important. In support, Wahlin reported that nurses need empowerment activities and that internal and external interventions affect psychological empowerment. Job satisfaction represents employees' general opinions and feelings about their jobs. According to a bibliometric analysis, the concept of empowerment in nurses has a strong and close relationship with job satisfaction.It has been determined that it has a positive impact. Employees who feel more confident and empowered in their ability to perform their jobs successfully tend to be more engaged in that job and experience greater job satisfaction. Psychological empowerment practices increase job satisfaction by positively influencing employees' belief that they are doing their jobs well, while also motivating employees to perform more successfully. Larrabee et al. emphasized that nurses who believe in their own abilities and do not focus on their shortcomings feel more empowered. Empowerment has many positive effects, such as greater productivity in nurses and better performance in nursing practice. Practices based on psychological empowerment principles increase the self-esteem, confidence, problem-solving skills, and innovative behaviors of healthcare professionals. In these respects, psychological empowerment programs can contribute to increasing nurses' job satisfaction. Innovative behavior refers to the process by which individuals develop, implement, and disseminate new ideas to create innovations in organizational processes. This behavior encompasses not only the generation of creative ideas for new products and technologies, but also the development of ideas for improving administrative procedures that contribute to strengthening social relationships in the workplace and increasing organizational efficiency. A meta-analysis conducted to examine the relationship between psychological empowerment and innovative work behavior indicated a strong effect size (r=0.580). Research on psychological empowerment interventions is still in its developmental stage and is quite limited. While several studies on the psychological empowerment of nurses exist in the literature, structured, long-term psychological empowerment programs appear to be limited. Examples of these programs include the online empowerment program for nurses developed by Bard et al.; "Huddling," developed by Im et al. to empower newly graduated nurses in Korea and increase their institutional commitment and resilience; an empowerment-based education program (EBEP) developed by Chang et al. for public health nurses in Taiwan; Özbaş and Tel's psychodrama-based psychological empowerment program for oncology nurses; Dirik and Seren's study, which aims to develop psychological empowerment by developing authentic leadership; and psychological support-based empowerment programs that focus on empowering nurses by providing them with direct psychological support. Existing interventions are generally based on traditional educational methods. The lack of studies using alternative and innovative methods, especially game-based educational programs, is noteworthy. Empowerment involves learning to take initiative and respond creatively to challenges encountered at work. Therefore, the empowerment process is viewed as a skill that can be learned and acquired through reinforcement. Group workshops and systematic educational programs are known to effectively increase psychological empowerment among nurses. Chang et al. stated that education-based psychological empowerment programs can increase the psychological empowerment of nurses. It is known that individuals can also be psychologically empowered through educational interventions. Games as an educational intervention are recognized for their effectiveness in improving cognitive and emotional learning. Games are also known to enhance creativity and innovative behavior. Games reinforce a sense of competence and achievement, while group workshops, including question-and-answer activities, group discussions, and sharing experiences within the group, allow participants to discover their own strengths and those of others. Developing psychological empowerment programs through training and programs that include games can help nurses create a fun space for themselves in busy work environments, boost their psychological strength, and increase their job satisfaction and innovative behaviors. Through games, nurses will have the opportunity to experience many practices such as collaboration and teamwork, role sharing, managing work, and completing work. Winning games can contribute to the success of the pros and cons.Solving the puzzle and being able to develop and implement different strategies will strengthen the sense of accomplishment, which will increase nurses' belief that they are effective in their work and help them experience job satisfaction. Feedback from other group members will also contribute to the psychological empowerment of participants.

Board games, also known as board games or box games, are games played by moving game pieces or checkers according to specific rules, usually on a flat surface or surfaces made of materials such as cardboard, wood, or plastic. Board games are characterized by gamified learning, where multiple players interact while playing with cards or checkers. A systematic review on the effectiveness of programs using board games indicated that board games improve knowledge understanding, interpersonal interaction, participatory learning, clinical reasoning, and cognitive functions. Board games can foster skills such as teamwork, empathy, and communication by fostering group interaction. These games can also help nurses develop strategies to cope with the challenges they face. It is also known that board games can increase clinical reasoning, problem-solving, and learning engagement in nurses. In the healthcare field, board games have generally focused on increasing anatomical knowledge, identifying high-risk medications for new nurses, their effects on patient cognitive function, and psychiatric care. Board games have become very popular and fun to play. However, each new game requires a special table and accessories. For these reasons, playing board games in a digital environment increases accessibility. The digitalization of board games is relatively new and has offered advantages such as ease of mass distribution, the convenience of group members gathering simultaneously, cost-effectiveness, and the ease of changing games without the need to physically produce new materials. Digital board games are known as digitized versions of traditional board games. These games are played on digital devices such as computers, tablets, or smartphones and typically offer multiplayer experiences online. Digital board games preserve the rules and mechanics of physical games while enriching the user experience with the advantages offered by digital platforms. Developments in the digital age, with many solutions such as mobile apps, games, software platforms, etc., make the use of digital board games considerably easier. The increasing variety of game options, in particular, has made digital board games a topic of considerable interest not only from an entertainment perspective but also from an academic perspective. Digital board games are used as effective tools in education and training. Furthermore, digital board games offer advantages such as increasing players' social interaction, enhancing problem-solving skills, and encouraging teamwork. Digital board games are almost universally prevalent across cultures and age groups. They are also receiving increasing attention from healthcare professionals due to their tremendous potential for education and therapy. With these characteristics, digital board games can be an effective tool in interventions designed to promote psychological empowerment, job satisfaction, and innovative behaviors, and were selected as the psychological empowerment intervention in our study.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 45 (although there are differing opinions in the literature on the age limit, the 45-year-old age limit encompasses a period when the effects of aging are more pronounced),
* Voluntarily participating in the study and having given written consent,
* Working a mix of day and night shifts (arrangements such as working only during the day, only at night, or with maternity leave will be excluded),
* Not receiving any other psychological training or therapy during the study dates,
* Not holding any additional job,
* Not participating in any additional program,
* Having at least one year of work experience,
* Not having a physical or mental illness that would prevent participation in the program,
* Having a bachelor's degree,
* Working as a nurse in the relevant institution during the study dates,
* Possessing and being able to use a computer, mobile phone, etc., to play digital games and participate in online group workshops and online training presentations.

Exclusion Criteria:

* Not meeting inclusion criteria

  • Exclusion criteria from the study:
* Failure to attend 2 or more sessions (attending less than 70% of the sessions),
* Withdrawal from the study voluntarily,
* Developing health problems that prevent participation after starting the program,
* Failure to complete all six sessions for various reasons (illness, moving, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Psychological Empowerment Level | Pre-intervention (baseline), post-intervention (week 6), 1-month follow-up, 3-month follow-up.
  Nurses' psychological empowerment levels will be assessed using the Psychological Empowerment Scale developed by Spreitzer. The scale's validity and reliability in Turkish were conducted by Üner & Turan. The scale consists of 12 items and uses a 7-point Likert-type scale (1 = strongly disagree, 7 = strongly agree). The minimum score is 12, and the maximum score is 84. Higher scores indicate higher levels of psychological empowerment.

SECONDARY OUTCOMES:
Job Satisfaction Level | Pre-intervention (baseline), post-intervention (week 6), 1-month follow-up, 3-month follow-up.
  Nurses' job satisfaction levels will be assessed using the Job Satisfaction Scale, developed by Brayfield and Rothe, abbreviated by Judge et al., and validated and verified in Turkish by Başol & Çömlekçi. The scale is a one-dimensional, five-item, 5-point Likert-type scale (1=Strongly disagree, 5=Strongly agree). The minimum score is 1, and the maximum score is 5. Higher scores indicate higher levels of job satisfaction.
Innovative Behavior Level | Pre-intervention (baseline), post-intervention (week 6), 1-month follow-up, 3-month follow-up.
  Description: Nurses' innovative behavior levels will be assessed using the Innovative Behavior Scale, developed by Scott and Bruce and validated and verified in Turkish by Çalışkan et al. The scale consists of six items and is a 5-point Likert-type scale (1 = Strongly disagree, 5 = Strongly agree). The minimum score is 6, and the maximum score is 30. Higher scores indicate higher levels of innovative behavior.

OTHER OUTCOMES:
Program Evaluation | Immediately after the intervention is completed (week 6).
  The intervention group's opinions on the program duration, content, method, and benefits will be collected using the Program Evaluation Form prepared by the researcher. The form includes three structured questions (e.g., duration of instruction, liking of board games) and an open-ended suggestion section. It is not a scored scale.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz KANTEK, Prof. Dr., Study Director — Akdeniz University

IPD SHARING:
Plan to Share IPD: Yes
When all the data collected are analyzed, that is, reported, it will form the basis of the results of a publication and will be stated as a doctoral thesis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2025 until October 2026
Access Criteria: They can access the study protocol and study purpose/description through this platform.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT07239882/Prot_SAP_ICF_000.pdf